CLINICAL TRIAL: NCT04271280
Title: Treatment of High and Very High riSk Dyslipidemic pAtients for the PreveNTion of CardiOvasculaR Events in Europe - a MultInatioNal ObservatIonal Study (SANTORINI)
Brief Title: Treatment of High and Very High riSk Dyslipidemic pAtients for the PreveNTion of CardiOvasculaR Events
Acronym: SANTORINI
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: DSE-HCL-01-19-EU
Record Dates: First submitted 2020-02-07; First posted 2020-02-17 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Dyslipidemia; Cardiovascular Diseases; Hypercholesterolemia; Atherosclerotic Cardiovascular Disease
Keywords: High-risk dyslipidemic; Low-density lipoprotein cholesterol; Cardiovascular disease; Lipid modifying therapies; Dyslipidemia; Hypercholesterolemia; Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Dyslipidemias; Cardiovascular Diseases; Hypercholesterolemia; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High Risk and Very High Risk Dyslipidemic Participants: Participants are classified as High and Very High Risk (as assessed by the Framingham risk score for High Risk participants and the SMART score for Very High Risk participants) as well as if previously or newly diagnosed.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — This is a non-interventional study.

SUMMARY:
High and Very High Risk cardiovascular patient journeys seems to vary from country to country, and current understanding of the process is incomplete. This real-life observational study which documents meaningful patient journey-related parameters can be expected to provide meaningful insight into the care process, country-by-country.

DETAILED DESCRIPTION:
Suffering from hypercholesterolemia is a major health concern in Europe. Appropriate medical treatment lowers low density lipoprotein cholesterol and reduces the incidence of clinical cardiovascular events. Despite the multiple available treatments, many patients remain inadequately treated or even untreated and some lipid-lowering drugs may be associated with an increase in events like side effects or increase in diabetes. As this is a non-interventional study, only data from routine clinical practice will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Very High Risk and High Risk dyslipidemic patients requiring LMTs
* Not simultaneously participating in any interventional study
* Providing written informed consent for participation in the study (Informed consent form)
* Life expectancy > 1 year

Exclusion Criteria:

* Not applicable; non-interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High risk and very high-risk participants requiring lipid-modifying therapies
Sampling Method: Non-Probability Sample
Enrollment: 9559 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Contact for Clinical Trial Information, Study Director — Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company
Locations (537):
- Austria (18):
  - Krankenhaus St. Josef Braunau GmbH, Braunau am Inn
  - LKH-Univ. Klinikum Graz, Graz
  - Medizinische Universität Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - KABEG Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Konventhospital der Barmherzigen Brüder Linz, Linz
  - Privatklinik Wehrle-Diakonissen, Salzburg
  - Ordination Universitätsdozent Dr. Alexander Kober, Sankt Aegyd am Neuwalde
  - Ordination Dr. med. univ. Evelyn Fließer-Görzer, Sankt Stefan
  - Ordination Dr. Thomas Maca / Evangelische KH Wien, Vienna
  - Ordination Dr. Thomas Maca / Evangelisches KH Wien, Vienna
  - Krankenhaus Rudolfstiftung, Vienna
  - Zentrum für Klinische Studien Dr. Hanusch GmbH, Vienna
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Ordination Dr. Reinhard Sock, Vienna
  - Krankenhaus Hietzing mit neurologischem Zentrum Rosenhügel, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf, Vienna
  - Internistische Facharztpraxis Frau Dr. Carmen Gelsinger, Zams
- Belgium (27):
  - ASZ, Aalst
  - Imeldaziekenhuis, Bonheiden
  - Clinique Saint-Luc, Bouge
  - AZ KLINA, Brasschaat
  - CHU Saint Pierre, Brussels
  - CHU Brugmann, Brussels
  - CUB Hospital Erasme, Brussels
  - UZ Brussel, Brussels
  - Cliniques de l'Europe, Brussels
  - Private practice, De Haan
  - Private practice, De Pinte
  - AZ Sint Blasius, Dendermonde
  - AZ Sint Lucas, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Cabinet de médecine générale, Gribomont
  - CH Jolimont-Lobbes, Haine-Saint-Paul
  - CHR de Huy, Huy
  - Jan Yperman Hospital, Ieper
  - AZ Groeninge VZW, Kortrijk
  - CHC Liège, Liège
  - AZ Delta, Roeselare
  - AZ Glorieux, Ronse
  - Sint Trudo, Sint-Truiden
  - Private practice, Tienen
  - BVBA Dr CAPIAU, Wetteren
  - CHU UCL Namur, Yvoir
  - Z Sint Elisabeth Zottegem, Zottegem
- Denmark (11):
  - Hjerteklinik Osterbro, Copenhagen
  - Amager Hospital, Copenhagen
  - Bispebjerg-Frederiksberg Hospital, Copenhagen
  - Bispebjerg/ Frederiksberg Hospital, Copenhagen
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Frederiksberg Hjerteklinik, Frederiksberg
  - Stroke center Rigshospitalet, Glostrup Municipality
  - Rigshospitalet (Copenhagen University Hospital) - Glostrup (Glostrup Hospital), Glostrup Municipality
  - Gentofte Hospital, Hellerup
  - Kobenhavns Universitet - Holbaek Sygehus, Holbæk
  - Slagelse sygehus, Slagelse
- Finland (24):
  - Mehiläinen Leppävaara, Espoo
  - Geri-Med Oy, Helsinki
  - Pihlajalinna Dextra, Helsinki
  - Pihlajalinna (Site 04-007), Joensuu
  - Pihlajalinna (Site 04-022), Joensuu
  - StudyCor Oy, Jyväskylä
  - Terveystalo Kalajoki, Kalajoki
  - Aava Kerava Medical Center, Kerava
  - Terveystalo Kokkola, Kokkola
  - Mehiläinen Kuopio, Kuopio
  - Lappeenrannan Työterveys - Site 4024, Lappeenranta
  - Lappeenrannan Työterveys - Site 4025, Lappeenranta
  - Terveystalo, Loimaa
  - Oulu University Hospital, Oulu
  - Satasairaala, Pori
  - Sastamalan seudun sosiaali- ja terveyspalvelut, Sastamala
  - Seinäjoki Central Hospital, Seinäjoki
  - Terveystalo Tampere, Tampere
  - Tampere University Hospital, Tampere
  - Mehiläinen Turku Kauppiaskatu, Turku
  - Turku University Hospital, Turku
  - Terveystalo Myyrmäki (Site 04015), Vantaa
  - Terveystalo Myyrmäki (Site 04017), Vantaa
  - Finla Työterveys Vantaa, Vantaa
- France (36):
  - 4 Rue Larrey, Angers
  - Cabinet médical Louis Blanc, Anzin
  - Clinique d'Argonay, Argonay
  - Hôpital Henri Duffaut, Avignon
  - Centre de Cardiologie et d'exploration de la Côte Basque, Bayonne
  - 151 rue Georges Clémenceau, Breteuil
  - 4 Rue du Capitaine Drillien, Chalon-sur-Saône
  - Centre Hospitalier de Chateauroux, Châteauroux
  - CH Compiègne, Compiègne
  - Centre Hopsitalier Alpes Leman, 552 Route de Findrol, Contamine-sur-Arve
  - 619 Rue de Saint Vaast, Flesselles
  - CHU Grenoble, Grenoble
  - 2 Boulevard Victor Hugo, Istres
  - 2 Rue du Dr Schweitzer, La Rochelle
  - Hôpital Louis Pasteur, Le Coudray
  - 222 Avenue du Mont Gaillard, Le Havre
  - Hôpital Marie Lannelongue, Le Plessis-Robinson
  - Institut Cœur Poumons, Boulevard du Pr Leclercq, Lille
  - Centre Hospitalier de Lisieux, 4 Rue Roger Aini, Lisieux
  - Centre Hospitalier La Timone, Marseille
  - Clinique de Meudon, Meudon-la-Forêt
  - Clinique du Pont de Chaume, Montauban
  - Clinique du Millénaire, Montpellier
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Hôpital Guillaume et René Laennec, Nantes
  - Centre Hospitalier de Nice, Nice
  - CHU Carémeau, Nîmes
  - Cabinet médical du docteur Cohen, Paris
  - Cabinet de cardiologie, Paris
  - Hôpital Pitié Salpétrière, Paris
  - Centre Hospitalier de Pau, Pau
  - Clinique Sant Hilaire, Rouen
  - 82 Avenue de Pontaillac, Royan
  - Hôpital Sainte Musse, Toulon
  - Centre Hospitalier Toulouse, Toulouse
  - Hôpital Guy Chatillez, Tourcoing
- Germany (139):
  - Downtown Clinic Aachen, Aachen
  - Kardiologische Praxis Aachen, Aachen
  - Praxis Delonge, Aachen
  - Kliniken an der Paar - Krankenhaus Aichach, Aichach
  - Oberpfalz Research GbR, Amberg
  - MVZ Aue, Aue
  - Kardiologische Praxis, Bad Elster
  - Kardiologische Praxis, Bad Homburg
  - Universitäts-Herz-Zentrum Freiburg-Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik Forschungsgesellschaft mbH, Bad Nauheim
  - Herz - u. Diabeteszentrum NRW, Bad Oeynhausen
  - Praxis am Landratspark, Bad Segeberg
  - Gemeinschaftspraxis für Herz und Lunge, Bamberg
  - Kardiologische Praxis, Bechhofen
  - Diabetespraxis Prenzlauer Allee, Berlin
  - Praxis Rankestraße, Berlin
  - MVZ Dres. Ramdohr - Praxis für Cardiovascular und Ultraschalldiagnostik, Berlin
  - Praxis Dr. Matthias Claus, Berlin
  - Kardiologische Facharztpraxis Dr. Anne Winkelmann, Berlin
  - Charité Campus Virchow, Berlin
  - Vivantes Humboldt-Klinikum, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Marienhaus-Klinikum Eifel Bitburg, Bitburg
  - Städtisches Klinikum Brandenburg, Brandenburg
  - Kardiologie an der Paulikirche, Braunschweig
  - Kardiologie im Friedrichspalast Bruchsal, Bruchsal
  - MediClin Reha-Zentrum Spreewald, Burg
  - MVZ am Küchwald, Chemnitz
  - Praxis Dipl.med Schermaul, Chemnitz
  - Kardiologische Praxis, Chemnitz
  - MVZ Polymed, Chemnitz
  - St. Josefs-Hospital Cloppenburg, Cloppenburg
  - Klinikum Coburg GmbH, Coburg
  - MVZ Gesundes Herz, Cologne
  - Praxis Dr. Menzel, Dessau
  - Klinikum Lippe GmbH, Detmold
  - Kardiologische Gemeinschaftspraxis, Dortmund
  - Sankt-Johannes-Hospital, Dortmund
  - Kardiologische Gemeinschaftspraxis Dres. Wetzel/Willgeroth, Dortmund
  - Zentrum für klinische Prüfungen in der Facharztzentrum Dresden-Neustadt GbR, Dresden
  - Praxis Dr. Methfessel, Dresden
  - Hausärztlich-Kardiologisches MVZ "Am Felsenkeller" GmbH, Dresden
  - Studienzentrum Dr. Faulmann, Dresden
  - Dres. Günther/Kolschmann, Dresden
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Praxis Dres. Jänsch/Varnai, Dresden
  - Praxis Dipl. - Med. Petra Herrmann - Fachärztin für Innere Medizin, Eisenach
  - Kardiologische Praxis, Elsterwerda
  - Elisabeth Krankenhaus Essen, Essen
  - Universitätsklinikum Essen, Essen
  - Medizentrum Essen Borbeck, Essen
  - Klinikum Frankfurt Hoechst GmbH, Frankfurt
  - MVZ Altstadt-Carree Fulda GmbH, Fulda
  - Evangelisches Krankenhaus Gelsenkirchen, Gelsenkirchen
  - Kardiologische Praxis, Gera
  - Kardiologische Praxis, Gotha
  - Praxis für Gefäßmedizin, Görlitz
  - Universitätsmedizin Göttingen, Göttingen
  - Praxis für Herzkreislauferkrankungen Greiz, Greiz
  - Evangelisches Krankenhaus Hagen-Haspe, Hagen
  - Gemeinschaftspraxis Dres. J. Hintze und M. Grundner, Hainstadt
  - Cardiologicum Hamburg-Wandsbek, Hamburg
  - Kardiologie am Tibarg, Hamburg
  - MVZ Prof. Detlef Mathey, Prof. Schofer GmbH, Hamburg
  - Kardiologische Praxis, Hanover
  - Kardiologische Praxis, Haßloch
  - Kardiologische Schwerpunktpraxis, Heidelberg
  - Praxis für Angiologie und Hämatologie, Heidelberg
  - Uniklinikum Heidelberg, Heidelberg
  - Praxis, Homburg
  - Kardiologie Oberschwaben - Bodensee Herz- und Gefäßpraxis, Isny
  - Kardiologische Praxis, Jena
  - Kardiopraxis Schirmer, Kaiserslautern
  - Kardiologie/Internistenteam Kamen, Kamen
  - SRH Klinikum Karlsbad-Langensteinbach, Karlsbach
  - B. Braun Ambulantes Herzzentrum MVZ GmbH, Kassel
  - CC Cleve-Studiencenter, Kleve
  - Studienzentrum der Inneren Medizin I & II am Klinikum Konstanz, Konstanz
  - Praxis für Innere Medizin / Kardiologie - Dr. med. E. Persicke / Dr. med. O. Scheuermann, Kornwestheim
  - Kardiologische Gemeinschaftspraxis, Leipzig
  - MediClin MVZ Leipzig, Leipzig
  - Praxis für Gefäßerkrankungen und Gerinnungsstörungen Leipzig, Leipzig
  - Gemeinschaftspraxis Dr. Täschner/Dr. Bonigut, Leipzig
  - MVZ Stoffwechselmedizin Leipzig, Leipzig
  - Universitätsklinikum Leipzig, Leipzig
  - Kardiologische Fachpraxis, Lengerich
  - Praxis Dr. med. Ilka Simon-Wagner, Lichtenfels
  - St. Vincenz-Krankenhaus, Limburg
  - Gemeinschaftspraxis Dr. Jens Biesenbaum und Dr. Uwe Gerbaulet, Löhne
  - Kardiologische Praxis Lohne, Löhne
  - Cardio Centrum Ludwigsburg-Bietigheim, Ludwigsburg
  - Kardiologische Praxisklinik Ludwigshafen, Ludwigshafen
  - Klinikum Lüdenscheid, Lüdenscheid
  - Dres. Erdmann/Schütz/Sicken, Lünen
  - St.Vincenz - u. Elisabeth-Hospital, Mainz
  - Universitätsklinikum Mainz Site 6186, Mainz
  - Universitätsklinikum Mainz Site 6187, Mainz
  - zero Praxen Mannheim, Mannheim
  - Universitätsklinikum Mannheim, Mannheim
  - Kardiologische Praxis, Markkleeberg
  - Praxis Dr. Ben-Chur, Meiningen
  - Kardiologie-Praxis, Moers
  - Gemeinschaftspraxis Dr. med. Martin Prohaska und Dr. med. Felix Schulte, Mühldorf
  - Herzquartier Mühlheim, Kardiologische Gemeinschaftspraxis Dres. med. A. Krapivsky & P. Kekes, Mühlheim
  - Zentrum für Diabetes und Gefäßerkrankungen Münster, Münster
  - Praxis für Innere Medizin, Münster
  - Universitätsklinikum Münster, Münster
  - Praxis für Innere Medizin und Angiologie, Nordhausen
  - Kardiologische Praxis Northeim, Northeim
  - Gemeinschaftspraxis Drs. Haggenmiller/Jeserich Kardiologie-Angiologie-Innere Medizin, Nuremberg
  - Kardiologie am Weißen Turm, Nuremberg
  - St. Vincenz-Krankenhaus GmbH, Paderborn
  - Kardiologische Praxis, Panitzsch
  - Kardiologische Praxis Papenburg (Site 6097), Papenburg
  - Kardiologische Praxis Papenburg (Site 6098), Papenburg
  - Kardiologische Praxis, Pirmasens
  - Cardiologicum Dresden/Pirna, Pirna
  - Kardiologie Potsdam, Potsdam
  - Kardiologische Gemeinschaftspraxis Potsdam, Potsdam
  - Paracelsus-Harz-Klinik Bad Suderode, Quedlinburg
  - Drs. Bauer/Buresch/Kösler, Regensburg
  - Gemeinschaftspraxis Herz Riesa, Riesa
  - Universitätsmedizin Rostock, Rostock
  - Zentrum für Prävention und Rehabilitation, Siegen
  - Kardiologische Praxis, Stahnsdorf
  - Praxis Dr. Birkenhagen, Stollberg
  - Drs. Knoebel @ Partner, Straubing
  - Praxis Dr. Michael Rother, Strausberg
  - Diabetologische Schwerpunktpraxis, Trier
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Studienzentrum der Herzklinik Ulm GbR, Ulm
  - Praxis Dr. Sabine Hansen, Unterwellenborn
  - Praxis für Prävention und Therapie, Villingen-Schwenningen
  - SHG Klinik Völklingen, Völklingen
  - GRN Klinik Weinheim, Weinheim
  - Forschungszentrum-Ruhr KliFoCenter GmbH, Witten
  - Klinikum Worms, Worms
  - Praxis Dr. Woitek, Wurzen
  - Praxis T. Schwarz, Zwenkau
- Ireland (7):
  - Beaumont Hospital, Beaumont, Dublin
  - Tramore Medical Clinic, Tramore, Waterford
  - Cork University Hospital, Cork
  - Mater Private Hospital, Dublin
  - St. James Hospital, Dublin
  - Beacon Hospital, Dublin
  - Turloughmore Health Centre, Galway
- Italy (85):
  - Ospedale Civile SS. Annunziata (MEDICINA INTERNA- DIPARTIMENTO DI MEDICINA E SCIENZE DELL'INVECCHIAMENTO), Chieti, Abruzzo
  - Ente Ecclesiastico Ospedale Generale Regionale "F.Miulli", Bari, Apulia
  - A.O.U. Consorziale - Policlinico Bari (Dipartimento di Medicina Interna), Bari, Apulia
  - A.O.U. Consorziale - Policlinico Bari, Bari, Apulia
  - A.O.U. Ospedali Riuniti, Foggia, Apulia
  - Presidio Ospedaliero Vito Fazzi, Lecce, Apulia
  - Azienda Ospedaliera Universitaria Mater Domini - Site 8042, Catanzaro, Calabria
  - Azienda Ospedaliera Universitaria Mater Domini - Site 8053, Catanzaro, Calabria
  - Azienda Ospedaliera Universitaria Mater Domini - Site 8059, Catanzaro, Calabria
  - Ospedale G. Jazzolino, Vibo Valentia, Calabria
  - A.O. San Giuseppe Moscati (U.O.C. Cardiologia/UTIC), Avellino, Campania
  - A.O. San Giuseppe Moscati, Avellino, Campania
  - A.O.R.N. San Pio - P.O. RUMMO, Benevento, Campania
  - Azienda Ospedaliera di Rilievo Nazionale(A.O.R.N.) "Sant'Anna e San Sebastiano" di Caserta, Caserta, Campania
  - Ospedale Civile Santa Maria Incoronata dell'Olmo, Cava de' Tirreni, Campania
  - A.O.R.N. Cardarelli, Napoli, Campania
  - A.O.R.N. Ospedale dei Colli, Napoli, Campania
  - A.O.U. FEDERICO II (U.O.C. Diabetologia), Napoli, Campania
  - A.O.U. Federico II, Napoli, Campania
  - A.O.U. "San Giovanni di Dio e Ruggi d'Aragona", Salerno, Campania
  - Ospedale Civile San Rocco, Sessa Aurunca, Campania
  - Ospedale di Bentivoglio, Bentivoglio, Emilia-Romagna
  - Ospedale Maggiore di Bologna, Bologna, Emilia-Romagna
  - A.O.U di Bologna-Policlinico S.Orsola-Malpighi (U.O. Medicina Interna), Bologna, Emilia-Romagna
  - Policlinico Sant'Orsola-Malpighi (U.O. Cardiologia), Bologna, Emilia-Romagna
  - Ospedale di Carpi, Carpi, Emilia-Romagna
  - Arcispedale Sant'Anna Ferrara (U.O. Cardiologia), Ferrara, Emilia-Romagna
  - Azienda Ospedaliera-Universitaria S. Anna di Ferrara (Dipartimento medico), Ferrara, Emilia-Romagna
  - A.O.U. Policlinico di Modena, Modena, Emilia-Romagna
  - Ospedale Civile di Baggiovara- AOU di Modena, Modena, Emilia-Romagna
  - Ospedale Unico della Valtidone, Piacenza, Emilia-Romagna
  - Ospedale Guglielmo da Saliceto, Piacenza, Emilia-Romagna
  - Arcispedale Santa Maria Nuova - Azienda USL/IRCCS Reggio Emilia, Reggio Emilia, Emilia-Romagna
  - Presidio Ospedaliero "Santa Maria della Misericordia" di Udine, Udine, Friuli
  - ASL Roma 6 - Ospedali Riuniti Anzio - Nettuno, Anzio, Lazio
  - Ospedale dei Castelli - ASL Roma 6, Rome, Lazio
  - Policlinico Universitario Campus Bio-Medico, Rome, Lazio
  - Policlinico Umberto I, Rome, Lazio
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio
  - Ospedale Policlinico Casilino, Rome, Lazio
  - Azienda Ospedaliera San Giovanni Addolorata, Rome, Lazio
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, Lombardy
  - ASST Spedali Civili P.O di Brescia, Brescia, Lombardy
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (U.O Medicina Generale 2), Brescia, Lombardy
  - Fondazione Poliambulanza Istituto Ospedaliero - Brescia, Brescia, Lombardy
  - IRCCS Multimedica, Milan, Lombardy
  - Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Centro Cardiologico Monzino - IRCCS (Unità Prevenzione dell'Aterosclerosi), Milan, Lombardy
  - Centro Cardiologico Monzino - IRCCS, Milan, Lombardy
  - Istituto Clinico Sant'Ambrogio, Milan, Lombardy
  - IRCCS Istituto Ortopedico Galeazzi, Milan, Lombardy
  - Grande Ospedale Metropolitano di Niguarda, Milan, Lombardy
  - Presidio ospedaliero Cardinal Massaia - A.S.L. AT (SOC Diabetologia e Malattie Metaboliche), Asti, Piedmont
  - Ospedale Regina Montis Regalis, Mondovì, Piedmont
  - Ospedale degli Infermi di Rivoli, Turin, Piedmont
  - A.O.U. Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Ospedale dei Castelli, Verbania, Piedmont
  - Ospedale Civile SS Annunziata (Dipartimento di Medicina Clinica e Sperimentale), Sassari, Sardinia
  - Ospedale Cannizzaro, Catania, Sicily
  - A.O.U. Policlinico "G. Martino" (U.O. Cardiologia), Messina, Sicily
  - Ospedale Buccheri La Ferla, Palermo, Sicily
  - Triolo Zancle Hospital, Palermo, Sicily
  - Ospedale Giovanni Paolo II, Ragusa, Sicily
  - INRCA -Ospedale U. Sestilli di Ancona, Ancona, The Marches
  - Ospedali Riuniti "Umberto I - Lancisi - Salesi, Ancona, The Marches
  - Ospedale Macerata, Macerata, The Marches
  - Ospedale di Bolzano (U.O. Cardiologia e Prove Funzionali), Bolzano, Trentino-Alto Adige
  - Ospedale San Giuseppe, Empoli, Tuscany
  - A.O.U. Careggi (S.O.D. Malattie Aterotrombotiche) - Site 8020, Florence, Tuscany
  - A.O.U. Careggi - Site 8041, Florence, Tuscany
  - A.O.U. Careggi - Site 8093, Florence, Tuscany
  - Ospedale S. Andrea - Usl Toscana Sud Est, Massa Marittima, Tuscany
  - Ospedale SS Cosma e Damiano di Pescia - Azienda Usl Toscana centro, Pescia, Tuscany
  - Università di Pisa, Pisa, Tuscany
  - Fondazione Toscana Gabriele Monasterio, Pisa, Tuscany
  - Ospedale Cisanello - A.U.O.P. Azienda Ospedaliera Universitaria Pisana, Pisa, Tuscany
  - Ospedale di Santo Stefano di Prato - Azienda Usl Toscana centro (UO di Cardiologia), Prato, Tuscany
  - Ospedale Santo Stefano di Prato - Azienda Usl Toscana Centro, Prato, Tuscany
  - Azienda Ospedaliero-Universitaria Senese Dipartimento Delle Scienze Mediche U.O.C. Medicina Interna e della Complessità, Siena, Tuscany
  - Ospedale Le Scotte, Siena, Tuscany
  - USL Umbria I, Perugia, Umbria
  - A.O. Santa Maria della Misericordia, Perugia, Umbria
  - Ospedale di Arzignano, Arzignano, Veneto
  - Ospedale Mater Salutis, Legnago, Veneto
  - Presidio Ospedaliero di Mirano - ULSS 3 Serenissima, Mirano, Veneto
- Netherlands (35):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Ziekenhuis Groep Twente (ZGT), Almelo
  - ZiekenhuisGroepTwente, Zilvermeeuw 1, Almelo
  - Meander Medical Center, Amersfoort
  - Meander Medisch Centrum, Maatweg 3, Amersfoort
  - Bovenij Zekenhuis, Amsterdam
  - Albert Schweitzerlaan 31, Apeldoorn
  - Gelre Ziekenhuis, Apeldoorn
  - Tergooi, Blaricum
  - Ijsselland Ziekenhuis, Prins Constanijnweg 2, Capelle aan den IJssel
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Reinier de Graafweg 5, Delft
  - Nico Bolkesteinlaan 75, Deventer
  - Van Weel Bethesda, Dirksland
  - Slingeland, Doetinchem
  - Gelderse Vallei, Ede
  - Medisch Spectrum Twente, Enschede
  - Admiraal de Ruijten Ziekenhuis, Goes
  - Groene Hart Gouda, Gouda
  - Boerhaavelaan 22, Haarlem
  - Ropcke Zweers hospital, Jan Weitkamplaan 4-a, Hardenberg
  - Saxenburgh Medisch Centrum, Hardenberg
  - Ziekenhuis St Jansdal, Harderwijk
  - Dr G.H. Amshoffweg 1, Hoogeveen
  - Treant Zorggroep, Hoogeveen
  - LUMC, Leiden
  - Ikazai Ziekenhuis, Rotterdam
  - Els Borst, The Hague
  - Rivierenland ziekenhuis Tiel, Tiel
  - ETZ, Tilburg
  - Nistelrodeseweg 10, Uden
  - University Medical Center Utrecht, Utrecht
  - Diakonessenhuis Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - Zaans Medisch Centrum, Zaandam
- Portugal (11):
  - Instituto do Coração, Carnaxide
  - Centro Hospitalar Universitario do Algarve, Faro
  - Associação Protetora de Diabéticos de Portugal, Lisbon
  - Hospital Egas Moniz (CHLO), Lisbon
  - Hospital Lusíadas de Lisboa, Lisboa, Lisbon
  - Centro Hospitalar Lisboa Norte - Site 10005, Lisbon
  - Centro Hospitalar Lisboa Norte - Site 10006, Lisbon
  - Clínica Cuida Mais, Mangualde
  - Centro Hospitalar Universitário São João (CHUSJ), Porto
  - Instituto CUF Porto, Porto
  - Centro Hospitalar de Entre Douro e Vouga, Santa Maria da Feira
- Spain (71):
  - Hospital de Alta Resolución de Sierra Norte, Constantina, Andalusia
  - H. Reina Sofia, Córdoba, Andalusia
  - Hospital de Alta Resolución de Ecija, Écija, Andalusia
  - H Juan Ramón Jiménez de Huelva, Huelva, Andalusia
  - H. Infanta Elena, Huelva, Andalusia
  - Centro Médico Puerto, Jerez de la Frontera, Andalusia
  - HG. Univ. De Jérez, Jerez de la Frontera, Andalusia
  - Hospital de Alta Resolución de Lebrija, Lebrija, Andalusia
  - H Carlos Haya, Málaga, Andalusia
  - H. Univ. Virgen Macarena, Seville, Andalusia
  - H. San Agustín, Seville, Andalusia
  - H. Alta Resolución de Utrera, Utrera, Andalusia
  - Hospital de Alta Resolución de La Janda, Vejer de la Frontera, Andalusia
  - H. San Eloy, Barakaldo, Basque Country
  - H. Univ. Basurto, Bilbao, Basque Country
  - H. Univ. de Basurto, Bilbao, Basque Country
  - Clinica Privada Orotava, La Orotava, Canary Islands
  - C S Colloto, Colloto, Castille and León
  - H Universitario De León, León, Castille and León
  - H Clínico de Salamanca, León, Castille and León
  - C S de la Alamedilla, Salamanca, Castille and León
  - H. General de Segovia, Segovia, Castille and León
  - Complejo Asistencial de Zamora, Zamora, Castille and León
  - H. Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - H de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - H. Universitari Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - Complejo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Complejo Hospitalario Univ. El Ferrol, Ferrol, Galicia
  - Complejo Hospitalario de Ourense, Ourense, Galicia
  - H. Clínico Univ. Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - H. Universitario Fuenlabrada, Fuenlabrada, Madrid
  - H. Univ. Infanta Sofía, San Sebastián de los Reyes, Madrid
  - H. Costa del Sol, Marbella, Málaga
  - H Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Fundación Alcorcón, Alcorcón
  - H. del Mar Site 11041, Barcelona
  - H. del Mar Site 11065, Barcelona
  - H. Univ. Basurto, Bilbao
  - Centro de Salud Colloto, Colloto
  - Hospital Univ. Getafe, Getafe
  - Hospital de Jerez, Jerez de la Frontera
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario de la Princesa Site 11054, Madrid
  - Hospital Universitario de la Princesa Site 11062, Madrid
  - Hospital Universitario de la Princesa Site 11075, Madrid
  - H Gregorio Marañon, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid
  - Clinica Universitaria de Navarra, Madrid
  - Clínica Universitaria de Navarra, Madrid
  - Fundación Jiménez Díaz, Madrid
  - H. Univ. Clínico San Carlos, Madrid
  - H. Univ. La Paz-Carlos III, Madrid
  - H. Universitario La Paz-Carlos III, Madrid
  - Hospital La Paz-Carlos III, Madrid
  - H. Univ. Ramón y Cajal, Madrid
  - H. Universitario 12 de octubre, Madrid
  - H. Clínico Virgen de la Arrixaca, Murcia
  - Complejo Hospitalario Universitario de Ourense (CHOU) Site 11003, Ourense
  - Complejo Hospitalario Universitario de Ourense (CHOU) Site 11052, Ourense
  - H. San Joan de Reus, Reus
  - Hospital Parc Tauli, Sabadell
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes
  - Hospital de Sant Joan Despí Moisès Broggi, Sant Joan Despí
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital General de Segovia, Segovia
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Sant Pau i Santa Tecla, Tarragona
  - Hospital HM de Torrelodones, Torrelodones
  - Centro de Salud Fuentes Norte, Zaragoza
- Sweden (11):
  - Falu Lasarett, Diab/Endo-mottagning, Falun
  - Sahlgrenska University Hospital, Gothenburg
  - Östra Sahlgrenska Universitetssjukhuset - Ostra Sjukhuse, Gothenburg
  - Värmdö Vårdcentral, Gustavsberg
  - Öbackakliniken, Härnösand
  - Länssjukhuset Ryhov, Jönköping
  - Capio Citykliniken, Lund
  - Skåne University Hospital, Malmo
  - Cityheart, Stockholm
  - Södersjukhuset Stockholm, Stockholm
  - Karolinska University Hospital, Huddinge, Stockholm
- Switzerland (11):
  - Kantonsspital Baden AG, Baden
  - Universitätsspital Basel, Basel
  - Hôpitaux Universitaires de Genève, Geneva
  - University of Lausanne Unisanté, Lausanne
  - Cardio Center Luzern, Lucerne
  - Kardiolab, Olten
  - Solothurner Spitäler AG, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Cardiologue FMH, Yverdon-les-Bains
  - Klinik Hirslanden, Zurich
  - Universitätsspital Zürich, Zurich
- United Kingdom (51):
  - Craigavon Area Hospital, Craigavon, Armagh
  - The Boathouse Sugery, Reading, Berkshire
  - Oak Tree Surgery, Liskeard, Cornwall
  - Newquay Health Centre, Newquay, Cornwall
  - The Alverton Practice, Penzance, Cornwall
  - Knowle House Surgery, Plymouth, Cornwall
  - Royal Cornwall Hospital, Truro, Cornwall
  - Carmel Medical Practice, Darlington, County Durham
  - Fellview Healthcare, Whitehaven, Cumbria
  - The Adam Practice, Poole, Dorset
  - Manor Park Medical Practice, Leicester, East Midlands
  - Southend University Hospital, Southend, Essex
  - Barts Health NHS Trust, London, Greater London
  - Church End Medical, London, Greater London
  - The Friarsgate Practice, Winchester, Hampshire
  - Burbage Surgery, Hinckley, Leicestershire
  - Liverpool Heart & Chest Hospital NHS Trust, Liverpool, Merseyside
  - Breckland Alliance, London, Norfolk
  - Carlisle Healthcare, Carlisle, North Cumbria
  - Pickering Medical Practice, Pickering, North Yorkshire
  - Whitby Group Practice, Whitby, North Yorkshire
  - Lakeside Surgery, Corby, Northamptonshire
  - Danes Camp Medical Centre, Northampton, Northamptonshire
  - Ormeau Clinical Trials Ltd, Belfast, Northern Ireland
  - Branch End Surgery, Stocksfield, Northumberland
  - Princess Royal Hospital, Shrewsbury, Shropshire
  - Princess Royal Hospital, Telford, Shropshire
  - Heart of Bath Medical Partnership, Bath, Somerset
  - Clifton Medical Centre, Rotherham, South Yorkshire
  - Brockwood Medical Practice, Brockham, Surrey
  - Staploe Medical Centre, Soham, Surrey
  - North Tyneside General Hospital, North Shields, Tyne and Wear
  - Sunderland Royal Hospital, Sunderland, Tyne and Wear
  - Glan Clwyd Hospital, Bodelwyddan, Wales
  - Sherbourne Medical Centre, Royal Leamington Spa, Warwickshire
  - Huddersfield Hospital, Swindon, West Yorkshire
  - Great Western Hospital Swindon, Huddersfield, Wiltshire
  - Great Western Hospital Swindon, Swindon, Wiltshire
  - Huddersfield Hospital, Huddersfield, Yorkshire
  - The Atherstone Surgery, Atherstone
  - Layton Medical Centre, Blackpool
  - Waterloo Medical Care, Blackpool
  - Llanedeyrn Health Centre, Cardiff
  - Ely Bridge Surgery, Cardiff
  - Holderness Health Surgery, Hedon
  - Hull Royal Infirmary, Hull
  - Temple Sowerby Medical Practice, Penrith
  - Wansford and Kings Cliffe Practice, Peterborough
  - Panthera Preston, Preston
  - Ecclesfield Group Practice, Sheffield
  - Royal Albert Edward Infirmary, Wigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arca M, Calabro P, Solini A, Pirillo A, Gambacurta R, Ray KK, Catapano AL; SANTORINI Italian Group. Challenges in achieving LDL-C goals: Insights from the Italian SANTORINI study cohort. Nutr Metab Cardiovasc Dis. 2026 Feb;36(2):104412. doi: 10.1016/j.numecd.2025.104412. Epub 2025 Oct 14. PMID 41125511
- [Derived] Mostaza JM, Garcia-Ortiz L, Suarez Tembra MA, Talavera Calle P, Chimeno Garcia J, Escolar Perez V, Diaz-Diaz JL, Manzano-Espinosa L, Catapano AL, Ray KK, Diaz Moya G, Pedro-Botet Montoya J; en representacion del grupo de investigadores de SANTORINI Espana. Failure of LDL-C goals achievement and underuse of lipid-lowering therapies in patients at high and very high cardiovascular risk: Spanish subset from the European SANTORINI study. Rev Clin Esp (Barc). 2025 Feb;225(2):78-84. doi: 10.1016/j.rceng.2024.11.004. Epub 2024 Nov 28. PMID 39613100
- [Derived] Ray KK, Haq I, Bilitou A, Manu MC, Burden A, Aguiar C, Arca M, Connolly DL, Eriksson M, Ferrieres J, Laufs U, Mostaza JM, Nanchen D, Rietzschel E, Strandberg T, Toplak H, Visseren FLJ, Catapano AL; SANTORINI Study Investigators. Treatment gaps in the implementation of LDL cholesterol control among high- and very high-risk patients in Europe between 2020 and 2021: the multinational observational SANTORINI study. Lancet Reg Health Eur. 2023 Apr 5;29:100624. doi: 10.1016/j.lanepe.2023.100624. eCollection 2023 Jun. PMID 37090089

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 9559 participants were documented in this study (all-documented patients set; APS). Of these 9559 participants, 11 failed screening and 5 were not included due to end of enrollment. A total of 9543 participants were included in the Baseline Analysis Set (BAS) at 580 centers in 14 countries. Of these 9543 participants, a total of 9136 were included in the Full Analysis Set (FAS).
Groups:
- High Risk and Very High Risk Dyslipidemic Participants: Participants were classified as High and Very High Risk (as assessed by the Framingham risk score for High Risk participants and the SMART score for Very High Risk participants) as well as if previously or newly diagnosed.
Period: Overall Study
Arm/Group | High Risk and Very High Risk Dyslipidemic Participants
Started | 9559
Baseline Analysis Set (The Baseline Analysis Set (BAS) consisted of all eligible patients of the All-Documented Patient Set (APS) for whom adequate baseline information was available.) | 9543
Full Analysis Set (The Full Analysis Set (FAS) consisted of all patients from the BAS with any available 1-year follow-up data (including study termination data where the reason for termination was death).) | 9136
Completed | 8954
Not Completed | 605
Not completed — Lost to Follow-up | 300
Not completed — Death | 153
Not completed — Withdrawal of consent by patient | 59
Not completed — Other | 51
Not completed — No end of study information | 42

BASELINE CHARACTERISTICS:
Population: Baseline demographic characteristics were assessed in the Baseline Analysis Set.
Arm/Group | High Risk and Very High Risk Dyslipidemic Participants
Number analyzed (Participants) | 9543
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2618
  Male | 6925
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 658
  Portugal | 120
  Switzerland | 169
  Spain | 1043
  Austria | 306
  Netherlands | 535
  Sweden | 192
  Belgium | 530
  Ireland | 100
  Finland | 338
  Denmark | 319
  Italy | 2089
  France | 855
  Germany | 2289

OUTCOME MEASURES:

1. Primary Outcome: Mean Low Density Lipid-Cholesterol (LDL-C) Levels in High and Very High Risk Cardiovascular Participants
Description: Blood plasma samples were used to assess LDL-C levels.
Time Frame: Baseline up to 12 months post-enrollment
Population: Low Density Lipid-Cholesterol (LDL-C) levels were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | High Risk and Very High Risk Dyslipidemic Participants
Number analyzed (Participants) | 8537
mmol/L
  Baseline | 2.40 (1.20)
  1 Year: number analyzed (Participants) | 7507
  1 Year | 1.99 (0.94)

2. Primary Outcome: Number of Participants Utilizing Any Treatment Modality to Manage Plasma Levels of Low Density Lipid-Cholesterol (LDL-C) in High and Very High Risk Participants Requiring Lipid Modifying Therapies (LMTs)
Description: Clinical events were assessed based on information captured in patient files/medical records.
Time Frame: Baseline up to 12 months post-enrollment
Population: Treatment modalities were assessed among participants requiring LMTs with available data in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk and Very High Risk Dyslipidemic Participants
Number analyzed (Participants) | 9136
Participants
  Received any LMT | 8931
  Received any statin | 7680
  Received any ezetimibe | 2538
  Received any other LMT | 2128

3. Secondary Outcome: Mean Atherosclerotic Cardiovascular Disease (ASCVD)-Modifying Cholesterol Fragment Levels in High Risk and Very High Risk Dyslipidemic Participants
Description: Blood plasma samples were used to assess ASCVD-modifying cholesterol fragment levels.
Time Frame: Baseline up to 12 months post-enrollment
Population: Mean ASCVD-modifying cholesterol levels were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | High Risk and Very High Risk Dyslipidemic Participants
Number analyzed (Participants) | 8531
mmol/L
  Baseline: HDL-C: number analyzed (Participants) | 8490
  Baseline: HDL-C | 1.27 (0.40)
  1 Year: HDL-C: number analyzed (Participants) | 7384
  1 Year: HDL-C | 1.28 (0.39)
  Baseline: Non-HDL-C: number analyzed (Participants) | 8428
  Baseline: Non-HDL-C | 3.02 (1.35)
  1 Year: Non-HDL-C: number analyzed (Participants) | 7339
  1 Year: Non-HDL-C | 2.58 (1.06)
  Baseline: Total Cholesterol | 4.31 (1.40)
  1 Year: Total Cholesterol: number analyzed (Participants) | 7457
  1 Year: Total Cholesterol | 3.86 (1.13)
  Baseline: Triglycerides: number analyzed (Participants) | 7841
  Baseline: Triglycerides | 1.70 (1.17)
  1 Year: Triglycerides: number analyzed (Participants) | 6664
  1 Year: Triglycerides | 1.56 (1.04)

4. Secondary Outcome: Mean Apolipoprotein B Levels in High Risk and Very High Risk Dyslipidemic Participants
Description: Blood plasma samples were used to assess Apolipoprotein B levels.
Time Frame: Baseline up to 12 months post-enrollment
Population: Mean apolipoprotein B levels were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | High Risk and Very High Risk Dyslipidemic Participants
Number analyzed (Participants) | 492
g/L
  Baseline | 0.92 (0.39)
  1 Year: number analyzed (Participants) | 458
  1 Year | 0.80 (0.34)

5. Secondary Outcome: Mean Lipid Protein A Levels in High Risk and Very High Risk Dyslipidemic Participants
Description: Blood plasma samples were used to assess lipid Protein A levels.
Time Frame: Baseline up to 12 months post-enrollment
Population: Mean lipid protein A levels were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High Risk and Very High Risk Dyslipidemic Participants
Number analyzed (Participants) | 882
mg/dL
  Baseline | 47.97 (53.87)
  1 Year: number analyzed (Participants) | 564
  1 Year | 51.24 (53.47)

6. Secondary Outcome: Mean Inflammatory High-Sensitive C-Reactive Protein (hsCRP) in High Risk and Very High Risk Dyslipidemic Participants
Description: Blood plasma samples were used to assess hsCRP levels.
Time Frame: Baseline up to 12 months post-enrollment
Population: Mean hsCRP levels were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | High Risk and Very High Risk Dyslipidemic Participants
Number analyzed (Participants) | 1818
mg/L
  Baseline | 6.90 (14.8)
  1 Year: number analyzed (Participants) | 1231
  1 Year | 4.3 (10.4)

7. Secondary Outcome: Number of Participants With Clinical Events Associated With Treatment Modalities, For Any LMT
Description: The safety outcome measure reports clinical events based on information captured in patient files/medical records. Participants may have reported more than one clinical event associated with any LMT.
Time Frame: Baseline up to 12 months post-enrollment
Population: Clinical events were assessed among participants requiring LMTs with available data in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk and Very High Risk Dyslipidemic Participants
Number analyzed (Participants) | 8931
Participants
  Patients with any clinical event associated with treatment modalities | 423
  Patients with muscle-associated symptoms | 338
  Patient with new-onset and/or worsening of diabetes mellitus | 2
  Patients with reduced kidney function | 19
  Patients with neurocognitive impairment | 8
  Patients with laboratory abnormality/abnormalities | 59
  Patients with missing event-type | 28
  Patients without any event | 8508

ADVERSE EVENTS:
Time Frame: Since this was a non-interventional study, adverse event and serious adverse event data were not collected. Standard ADR reporting followed regulations for the post-marketing setting. Figures on ADR are not reported here. Death was assessed from study baseline up to 12 months post-enrollment and is reported.
Description: Death data are reported from the Full Analysis Set (FAS) that consisted of all patients from the Baseline Analysis Set (BAS) with any available follow-up data.
Groups:
- High Risk and Very High Risk Dyslipidemic Participants: Participants were stratified as High and Very High Risk (as assessed by the Framingham risk score for High Risk participants and the SMART score for Very High Risk participants) as well as if previously or newly diagnosed.
Arm/Group | High Risk and Very High Risk Dyslipidemic Participants
All-Cause Mortality (participants affected / at risk) | 153/9136
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Medication selection and adherence, lifestyle and other risk factors were decided on by routine care and patient choices, leading to potential bias: a selection bias of the included patients, an information bias on data collected, and a confounding bias in the treatment administration. In the current analysis, all eligible patients were included and no specific methods were employed to minimize bias or confounding effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT04271280/Prot_SAP_000.pdf